CLINICAL TRIAL: NCT02116829
Title: Is There Room for Butter in a Healthy Diet? - A Randomized Controlled Dietary Human Intervention
Brief Title: Is There Room for Butter in a Healthy Diet?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A309
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Butter; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Danish butter, dairy (Experimental)
  Interventions: Other: Danish butter
- Olive oil, refined (Active Comparator)
  Interventions: Other: Olive oil

INTERVENTIONS:
Other: Danish butter — The effect of butter intake versus olive oil (refined) intake on blood lipids (primarily)
  Other Names: butter, diary
  Arms: Danish butter, dairy
Other: Olive oil
  Arms: Olive oil, refined

SUMMARY:
The aim of this study is to examine the effects in humans of a moderate butter intake on risk markers of cardiovascular disease compared to a diet with the same amount of olive oil (refined and therefore without polyfenols).

The primary parameters are total cholesterol, LDL- and HDL cholesterol and triglycerides. The secondary parameters are risk markers of diabetes type 2; plasma glucose and insuling as well as the inflammatory marker hs-CRP.

ELIGIBILITY:
Inclusion Criteria:

* Sign written consent
* Age: 20-70 y
* BMI: 18.5 - 32 kg/m2
* Healthy men and women (with no known diseases)

Exclusion criteria

* Current or previously cardiovascular disease, high blood pressure
* Diabetes Mellitus or other severe chronic disease, including severe allergies
* Use of dietary supplements and blood donations prior to, and during the study
* Known or suspected abuse of alcohol, drugs or medication
* Pregnant or are planning pregnancy during the study period
* Extreme physical activity level (more than 10 hours tough physical activity pr. week)
* Participation in other research studies
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the study staff

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | 5 weeks
LDL cholesterol | 5 weeks
HDL cholesterol | 5 weeks
Triglycerides | 5 weeks

SECONDARY OUTCOMES:
Insulin | 5 weeks
Glucose | 5 weeks
hs-CRP | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tine Tholstrup, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Engel S, Tholstrup T. Butter increased total and LDL cholesterol compared with olive oil but resulted in higher HDL cholesterol compared with a habitual diet. Am J Clin Nutr. 2015 Aug;102(2):309-15. doi: 10.3945/ajcn.115.112227. Epub 2015 Jul 1. PMID 26135349